CLINICAL TRIAL: NCT03271684
Title: The Effectiveness of the Adapted Bridge's Self-management Programme in South African Community-dwelling Stroke Survivors: A Randomized Controlled Trial
Brief Title: The Effectiveness of the Adapted Bridge's Self-management Programme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of the Western Cape (Other)
Responsible Party: Principal Investigator, Reham Nasir, Principal investigator, University of the Western Cape
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM17/2/7
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Self-Care; Self Efficacy
Keywords: stroke, self-management, Bridges, participation, function, self-efficacy
MeSH Terms: conditions — Stroke | interventions — Self-Management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blinded, participant and assessor blinded, randomised trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Will receive one session of up to one-hour per week over a six-week period in self-management in addition to their usual rehabilitation and workbook.
  Interventions: Other: self-management
- control group (Other): Will receive booklet consist of home exercises and education besides the usual care
  Interventions: Other: Control

INTERVENTIONS:
Other: self-management — one session of up to one-hour per week over a six-week period in addition to their usual rehabilitation. During each session strategies will be used to promote specific behaviors that exemplify the hallmarks of self-management. These behaviors include enabling patients to work out ways of taking control of their daily lives by setting small targets, recording their progress and problem-solving. The content of the sessions is determined by the patient and their personal goals rather than being professionally directed
  Arms: intervention group
Other: Control — Participants will receive usual rehabilitation treatment, they will also be given a booklet with education program and exercises they can perform at home.
  Arms: control group

SUMMARY:
The effectiveness of the adapted Bridge's self-management programme in South African community-dwelling stroke survivors: A randomized controlled trial with two arms will be used, with the intervention group receiving self-management sessions delivered by experienced therapists and usual care and control group will only receive usual care which includes a information booklet.

DETAILED DESCRIPTION:
This study aim to determine the effectiveness of the Adapted bridges self-management intervention on South African stroke patients' functional activity, self-efficacy, and participation. Method: This experimental study will make use of a randomized controlled design (RCT), consisting of one hundred and sixty eight stroke survivors recruited from different health care facilities within the Cape Metropolitan area. The study participants will be divided randomly into two groups, with one receiving the intervention - the experimental group - and the other receiving an educational booklet - the control group. Participants will be assessed at baseline, immediately post-intervention (six weeks), three and sixth-month post intervention, using standardized outcome measures (both subjective outcome measures and objective clinical tools). Ethical clearance and permission to conduct the study will be obtained and patient information will be kept confidential. Analyses will be conducted using descriptive statistics of frequencies and percentages for categorical variables and mean and standard deviation for continuous variables. Given the assumptions of equal variance, a two-way full factorial ANOVA will be computed in order to assess interaction between groups and intervention type.

ELIGIBILITY:
Inclusion Criteria:

* having a first ever stroke, by a physician, based on the WHO (1988) definition of stroke which is "rapidly developing clinical signs of focal (or global) disturbance of cerebral function, with symptoms lasting 24 hours or longer or leading to death, with no apparent cause other than of vascular origin"; ≥18 years of age; of sufficient cognition to participate: having a score of ≥24 points on mini-mental state examination (placing participants at matched mental status) ; are medically stable and; and are within the sub-acute to chronic phase of their rehabilitation (10 weeks to 6-months post stroke).

Exclusion Criteria:

* Participants will be excluded if they have serious medical conditions such as HIV/AIDS or TB, which could additionally affect the outcomes evaluated in this study. Participants with depression, having recurrent stroke, still receiving in inpatient rehabilitation, with cognitive or receptive language difficulties and are unable to comprehend the intervention will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Stroke Self-Efficacy Questionnaire(SSEQ): | baseline to the 6 months after intervention
  The SSEQ is a 13 point questionnaire developed by Jones et al (2008) and is aimed to determine the individuals perceived level of self-efficacy in completing a range of relevant functional tasks, such as walking, getting comfortable in bed, as well as several self-management tasks

SECONDARY OUTCOMES:
The Rivermead Mobility Index: | baseline to the 6 months after intervention
  is a 15 point index with various topics and questions aimed at objectively determining the participant's mobility level. According to Lennon & Johnson (2000) highly reliable between raters (ICC = 0.98, p < 0.001) with high internal consistency (Cronbach's alpha = 0.93).
Rivermead Activities of Daily Living Scale: | baseline to the 6 months after intervention
  is a 31 point scale used to determine the level of independence a participant has with self-care and household tasks of varying difficulty. It has an excellent overall test-retest reliability (ICC = 0.96) (Chen et al, 2007) and an excellent concurrent validity at 180 days post stroke (r = 0.93) (Hsueh et al, 2003).
The Mini-BESTest: | baseline to the 6 months after intervention
  is a 14-item clinical test that covers four components of balance control (anticipatory postural adjustments, postural responses, sensory orientation and stability in gait). Each item is scored from 0 (unable or requiring help) to 2 (normal) and the maximal score is 28 points. The Mini-BESTest has an excellent test-retest reliability (ICC = 0.96), with an excellent convergent validity (r = 0.96) (Godi et al, 2013).
The Subjective Index of Physical and Social Outcome scale | baseline to the 6 months after intervention
  a 10 point rating index aimed at determining the participants' perceived extent of participation within the community, with its main domains as perceived functioning and social connectedness. SIPSO has been shown to present an excellent test-retest reliability with ICC = 0.96 and has indicated a proven validity (Trigg & Wood, 2003).
National Institute for Health Stroke Scale | baseline to the 6 months after intervention
  is a 15 item neurologic examination that provides a quantitative measure of stroke-related neurologic deficit. According to Kasner et al, (1999) reliability Agreement between pairs of raters was also very good to excellent, with ICCs ranging from 0.70 to 0.89.
Action Research Arm Test | baseline to the 6 months after intervention
  is a 19 item scale divided into four subscales: grasp, grip, pinch, and gross movement. The items within each subscale are arranged on a 4-point ordinal scale ranging from 0 to 3, with 3 indicating normal performance on each item. The maximum score on the ARAT is 57 points According to McDonnell, 2008 Inter-rater and retest reliability have been shown to be high (ICC > 0.98) in studies involving patients with stroke and Concurrent validity has been confirmed by comparison with the upper limb component of the Fugl- Meyer Assessment and the Motor Assessment Scale (MAS).
6-minute walk test | baseline to the 6 months after intervention
  Functional ability will be assessed using the 6-minute walk test (6-MWT), a reliable and valid measure for the stroke population. Participants will be instructed to walk at a comfortable pace on a 30-m measured walkway for 6 minutes. The outcome will be the total distance covered during testing. 6MWT exhibits excellent test-retest reliability (ICC = 0.973; 95 % CI = 0.925 to 0.988), it presents a minimal detectable change of 54.1 m, and an acceptable concurrent validity (r = 0.52 to 0.89) (Fulk et al, 2008).

IPD SHARING:
Plan to Share IPD: Undecided
Currently not allowed by ethic to share the data with other researchers

REFERENCES:
- [Background] Jones F, Partridge C, Reid F. The Stroke Self-Efficacy Questionnaire: measuring individual confidence in functional performance after stroke. J Clin Nurs. 2008 Apr;17(7B):244-52. doi: 10.1111/j.1365-2702.2008.02333.x. PMID 18578800
- [Background] Lennon S, Johnson L. The modified rivermead mobility index: validity and reliability. Disabil Rehabil. 2000 Dec 15;22(18):833-9. doi: 10.1080/09638280050207884. PMID 11197520
- [Background] Chen HM, Hsieh CL, Sing Kai Lo, Liaw LJ, Chen SM, Lin JH. The test-retest reliability of 2 mobility performance tests in patients with chronic stroke. Neurorehabil Neural Repair. 2007 Jul-Aug;21(4):347-52. doi: 10.1177/1545968306297864. Epub 2007 Mar 12. PMID 17353463
- [Background] Hsueh IP, Wang CH, Sheu CF, Hsieh CL. Comparison of psychometric properties of three mobility measures for patients with stroke. Stroke. 2003 Jul;34(7):1741-5. doi: 10.1161/01.STR.0000075295.45185.D4. Epub 2003 May 29. PMID 12775883
- [Background] Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther. 2013 Feb;93(2):158-67. doi: 10.2522/ptj.20120171. Epub 2012 Sep 27. PMID 23023812
- [Background] Trigg R, Wood VA. The Subjective Index of Physical and Social Outcome (SIPSO): a new measure for use with stroke patients. Clin Rehabil. 2000 Jun;14(3):288-99. doi: 10.1191/026921500678119607. PMID 10868724
- [Background] Kasner SE, Chalela JA, Luciano JM, Cucchiara BL, Raps EC, McGarvey ML, Conroy MB, Localio AR. Reliability and validity of estimating the NIH stroke scale score from medical records. Stroke. 1999 Aug;30(8):1534-7. doi: 10.1161/01.str.30.8.1534. PMID 10436096
- [Background] McDonnell M. Action research arm test. Aust J Physiother. 2008;54(3):220. doi: 10.1016/s0004-9514(08)70034-5. No abstract available. PMID 18833688
- [Background] The World Health Organization MONICA Project (monitoring trends and determinants in cardiovascular disease): a major international collaboration. WHO MONICA Project Principal Investigators. J Clin Epidemiol. 1988;41(2):105-14. doi: 10.1016/0895-4356(88)90084-4. PMID 3335877
- [Background] Fulk GD, Echternach JL, Nof L, O'Sullivan S. Clinometric properties of the six-minute walk test in individuals undergoing rehabilitation poststroke. Physiother Theory Pract. 2008 May-Jun;24(3):195-204. doi: 10.1080/09593980701588284. PMID 18569856